CLINICAL TRIAL: NCT04861350
Title: Restoration of Lumbopelvic Movement Control: Effect of Injury History, and the Role of Cortical Control and Its Practical Application(2)
Brief Title: Lumbopelvic Movement Control: Effect of Injury History, and the Role of Cortical Control and Its Practical Application 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Yi-Fen Shih, Professor, National Yang Ming Chiao Tung University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YM110027E(2)
Record Dates: First submitted 2021-04-13; First posted 2021-04-27 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Biomechanical Phenomena
Keywords: motor control; imagery training; corticomuscular coherence; event-related synchronization/ desynchronization
MeSH Terms: interventions — Physical Conditioning, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- motor imagery with action observation (Experimental): The subjects will perform the exercises mentally for 3 sets with video, 10 reps for 1 set.
  Interventions: Other: motor imagery with action observation
- physical training (Experimental): The subjects will perform the exercise physically for 3 sets with supervision of investigator, 10 reps for 1 set.
  Interventions: Other: physical training
- combine physical training and motor imagery with action observation (Experimental): The subjects will perform the exercise mentally with video for 1 set and physically with supervision of investigator for 2 sets, 3 sets totally, 10 reps for 1 set.
  Interventions: Other: combine physical training and motor imagery with action observation

INTERVENTIONS:
Other: motor imagery with action observation — Standing clamshell exercise with elastic band, sliding, and Romanian deadlift exercise will be instructed to the subjects with video, and they will practice each exercise for 3 times in physical to familiarize with the program. Then, the subjects will mentally simulate each exercise with video 10 times for a set, 3 sets totally. With 2 min interval between each sets, it will take approximately 8 minutes to finish each movement. It will also take 3 min for resting between each program.
  Arms: motor imagery with action observation
Other: physical training — Standing clamshell exercise with elastic band, sliding, and Romanian deadlift exercise will be instructed to the subjects with video, and they will practice each exercise for 3 times in physical to familiarize with the program. Then, the subjects will physically perform each exercise with supervision of investigator 10 times for a set, 3 sets totally. With 2 min interval between each sets, it will take approximately 8 minutes to finish each movement. It will also take 3 min for resting between each program.
  Arms: physical training
Other: combine physical training and motor imagery with action observation — Standing clamshell exercise with elastic band, sliding, and Romanian deadlift exercise will be instructed to the subjects with video, and they will practice each exercise for 3 times in physical to familiarize with the program. Then, each exercises will be mentally simulated with video for a set and physically performed with supervision of investigator for 2 sets, 10 times for each set and 3 sets totally. With 2 min interval between each sets, it will take approximately 8 minutes to finish each movement. It will also take 3 min for resting between each program.
  Arms: combine physical training and motor imagery with action observation

SUMMARY:
Hip motor control ability is an important parameter for preventing sport injuries in lower limbs, and the training of hip motor control can enhance the lower extremity movement performance. Previous studies have demonstrated the benefits of motor imagery with action observation (AOMI) on motor control and muscle strength improvements, which also revealed that AOMI combined with physical training (AOMI-PT) can lead to better outcomes than physical training (PT) alone. Besides, monitoring the neurophysiological changes of brain activation and the functional connection to the peripheral muscular activation after training helps to understanding the mechanisms on the training effects.

Therefore, the aim of this study is to compare (1) the cortical control mechanisms between 3 types of motor control training strategies; and (2) the effects of 3 types of motor control training on hip motor control performance in healthy subjects.

DETAILED DESCRIPTION:
Hip motor control ability is an important parameter for preventing sport injuries in lower limbs, and the training of hip motor control can enhance the lower extremity movement performance. Previous studies have demonstrated the benefits of motor imagery with action observation (AOMI) on motor control and muscle strength improvements, which also revealed that AOMI combined with physical training (AOMI-PT) can lead to better outcomes than physical training (PT) alone. Besides, monitoring the neurophysiological changes of brain activation and the functional connection to the peripheral muscular activation after training helps to understanding the mechanisms on the training effects.

Therefore, the aim of this study is to compare (1) the cortical control mechanisms between 3 types of motor control training strategies; and (2) the effects of 3 types of motor control training on hip motor control performance in healthy subjects.

The investigators will recruit 45 healthy subjects and compare the effect of three types of motor control training (physical training, motor imagery with action observation, physical training combined motor imagery with action observation) on Y balance test performance, cortico-muscular coherence (CMC), and task-related spectral power (TRSP) changes. Due to only few studies about the issue, we will recruit extra 15 healthy athletes for pilot study to investigate the reliability of the research measurements and refine the protocols.

Chi squared test is used to examine the group differences such as gender, dominant side and activity level. The 2-way mixed analysis of variance (ANOVA) will be used to compare the intervention effect on motor control test and CMC between groups. One-way repeated measures ANOVA will be used to investigate the neurophysiological changes on brain activation during AOMI training, and the changes of AOMI-PT and PT group will be compared by independent t-test. The alpha level was set at 0.05.

ELIGIBILITY:
Inclusion Criteria:

* without pain or symptoms on lower extremities or spine which affects on daily activities or sports participants lasting for more than 1 week within 6 months.

Exclusion Criteria:

* any symptoms or surgery history on lumbar or lower extremities in the past 6 months and still interrupt daily activities or sports participants.
* any neurological or psychosocial disease affects on motor imagery ability.
* with drug or alcohol abuse history.
* with visual or vestibular abnormalities without correction, or with concussion history within 3 month

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2023-01-10 (Actual)

PRIMARY OUTCOMES:
Motor control ability | pre-intervention
  The subjects will stand on Y-balance kit with their dominant leg and reach their non-dominant legs to anterior, posterolateral and posteromedial direction following the tempo with 5 sec forward and 5 sec backward in sequence. The subjects will practice 4 times first to familiarize the test procedure, then the final three measurements were collected and normalized with subjects' lower limb length for statistical analysis.
Cortico-muscular coherence | pre-intervention
  The investigator will place 64-leads EEG on subjects' head and bipolar surface EMG(MP150, BIONOMADIX; BIOPAC, Systems, Inc.) on subjects' internal oblique abdominis, gluteus medius, gluteal maximus and adductor longus. The investigator will collect the signals and process them into cortico-muscular coherence as the functional connection between cortex and muscle during motor control task.
Task-related spectral power | immediately after the intervention
  The investigator will collect the EEG signals from subjects during the intervention, and the signals will be band-pass filtered (3-60 Hz) and processed with power spectrum density analysis to calculate frequency power at alpha (8-12 Hz) and beta (13-30 Hz) bands. The training data will be normalized with resting values to determine task-related synchronization or desynchronization, which represent the cortical activation changes during training.
Motor control ability | immediately after the intervention
  The subjects will stand on Y-balance kit with their dominant leg and reach their non-dominant legs to anterior, posterolateral and posteromedial direction following the tempo with 5 sec forward and 5 sec backward in sequence. The subjects will practice 4 times first to familiarize the test procedure, then the final three measurements were collected and normalized with subjects' lower limb length for statistical analysis.
Cortico-muscular coherence | immediately after the intervention
  The investigator will place 64-leads EEG on subjects' head and bipolar surface EMG(MP150, BIONOMADIX; BIOPAC, Systems, Inc.) on subjects' internal oblique abdominis, gluteus medius, gluteal maximus and adductor longus. The investigator will collect the signals and process them into cortico-muscular coherence as the functional connection between cortex and muscle during motor control task.

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Fen Shih, Ph.D, Study Director — Department of Physical Therapy and Assistive Technology, National Yang-Ming Chiao-Tung University
Locations (1):
- National Yang Ming University, Taipei, Taiwan